CLINICAL TRIAL: NCT02937376
Title: Effects of N-acetyl Cystein (NAC) Supplementation in G6PD Deficient Individuals After Acute Exercise
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTH_G6PD 2
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: G6PD Deficiency
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency | interventions — ethofenprox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetyl Cystein (Experimental): NAC supplementation (10 mg/kg/day) for 4 weeks in a counterbalanced manner to 12 G6PD deficient individuals.
  Interventions: Drug: N-acetyl cystein
- Placebo (Placebo Comparator): Placebo administration for 4 weeks in a counterbalanced manner to 12 G6PD deficient individuals.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-acetyl cystein — A trial of exercise before and after 4 weeks of N-acetyl cystein (NAC) supplementation.
  Other Names: Trebon
  Arms: N-acetyl Cystein
Other: Placebo — A trial of exercise before and after 4 weeks of placebo administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of N-acetyl Cystein (NAC) supplementation on redox status, physiological and biochemical parameters in G6PD deficient individuals after acute exercise.

DETAILED DESCRIPTION:
In a randomized double-blind, crossover design, 12 adult volunteers with G6PD deficiency of both sexes will be supplemented with either 10 mg/kg of NAC (experimental condition - EC) or placebo (control condition - CC) every day for 4 weeks. Before intervention, all participants will be informed about the study protocol, fill a medical history questionnaire and sign an informed consent form. Moreover, measurements of anthropometric characteristics and physiological parameters, as well as a VO2max test will be performed.

Participants will perform 4 trials of exercise (70% VO2max for 45min and 90% till exhaustion) before and after each condition. Blood samples will be collected before, immediately after and 1 hour after exercise. Moreover, measurements of anthropometric characteristics and physiological parameters will be performed before and after each condition. There will be a washout period of at 4 weeks between conditions.

ELIGIBILITY:
Inclusion Criteria:

* G6PD deficiency

Exclusion Criteria:

* Any uncontrolled health condition for which exercise is contraindicated
* Current use of dietary supplements or drugs
* Pregnant, pregnancy intention or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in redox status after exercise | Before, immediately after and 1 hour after each trial of exercise
  Indices of blood redox status

SECONDARY OUTCOMES:
Body composition | Before and after 4 weeks of NAC supplementation, before and after 4 weeks of placebo
  Body fat percentage
Blood pressure | Before and after 4 weeks of NAC supplementation, before and after 4 weeks of placebo
  Blood pressure at rest

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z Jamurtas, PhD, Study Director — University of Thessaly
Locations (1):
- Department of Physical Education & Sport Science of the University of Thessaly, Trikala, Karyes, Greece

REFERENCES:
- [Background] Georgakouli K, Deli CK, Zalavras A, Fatouros IG, Kouretas D, Koutedakis Y, Jamurtas AZ. Alpha-lipoic acid supplementation up-regulates antioxidant capacity in adults with G6PD deficiency. Food Chem Toxicol. 2013 Nov;61:69-73. doi: 10.1016/j.fct.2013.01.055. Epub 2013 Feb 14. PMID 23416142